CLINICAL TRIAL: NCT01579305
Title: Safety and Effectiveness of Juvéderm® Volbella With Lidocaine Versus Restylane-L® for Lip Volume Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan Medical (Industry)
Responsible Party: Sponsor
Organization: Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S15L-003
Record Dates: First submitted 2012-04-16; First posted 2012-04-17 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Lip Volume Enhancement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Juvéderm® Volbella with Lidocaine (Experimental): Subjects injected with Juvéderm® Volbella with Lidocaine in their lips
  Interventions: Device: Juvéderm® Volbella with Lidocaine
- Restylane-L® (Active Comparator): Subjects injected with Restylane-L® in their lips
  Interventions: Device: Restylane-L®

INTERVENTIONS:
Device: Juvéderm® Volbella with Lidocaine — Up to 4.0 mL at the discretion of the Investigator to achieve optimal results
  Arms: Juvéderm® Volbella with Lidocaine
Device: Restylane-L® — Up to 4.0 mL at the discretion of the Investigator to achieve optimal results
  Arms: Restylane-L®

SUMMARY:
The purpose of this study is evaluate lip fullness 3 months following treatment with Juvéderm® Volbella with Lidocaine or Restylane-L®

ELIGIBILITY:
Inclusion Criteria:

1. Desire enhancement of his/her vermilion borders and/or vermilion mucosa
2. Have a baseline score of Minimal or Mild, as assessed by the Investigator, according to the 5-point LFS (Minimal, Mild, Moderate, Marked, Very Marked)
3. Have established a realistic Lip Fullness treatment goal that the Investigator agrees is achievable

Exclusion Criteria:

1. Have undergone cosmetic facial, lip or perioral procedures [e.g., face-lift, or other surgeries, which may alter the appearance of the lips or perioral area (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, or other ablative procedures), tissue augmentation with dermal fillers or fat injections, or mesotherapy] anywhere in the face or neck, or Botox® Cosmetic injections in the lower face (below the orbital rim), within 6 months prior to entry in the study or be planning to undergo any of these procedures at any time during the study. NOTE: Prior treatment with HA fillers and/or collagen is allowed, provided the treatment was administered more than 6 months prior to study entry
2. Have ever received semi-permanent fillers or permanent facial implants, e.g., calcium hydroxyapatite, L-polylactic acid, polymethylmethacrylate (PMMA), silicone, expanded polytetrafluoroethylene (ePTFE) anywhere in the lips, or be planning to be implanted with any of these products at any time during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Cannes, France
- Glasgow, United Kingdom

REFERENCES:
- [Background] Raspaldo H, Chantrey J, Belhaouari L, Saleh R, Murphy DK. Juvederm volbella with lidocaine for lip and perioral enhancement: a prospective, randomized, controlled trial. Plast Reconstr Surg Glob Open. 2015 Apr 7;3(3):e321. doi: 10.1097/GOX.0000000000000266. eCollection 2015 Mar. PMID 25878932

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was defined as having signed the IRB-approved Informed Consent Form. Prior to randomization, 4 subjects were excluded as screen fails, leaving an "Intent-to-Treat" population of 281 subjects.
Period: Overall Study
Arm/Group | Subject Randomized to Receive VOLBELLA® | Subjects Randomized to Receive Restylane-L®
Started | 139 (Subjects that signed Informed Consent, passed screening criteria, and were randomized.) | 142 (Subjects that signed Informed Consent, passed screening criteria, and were randomized.)
Discontinued Before Treatment | 0 | 1
Continued After Treatment | 139 | 141
Completed | 118 | 115
Not Completed | 21 | 27

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are based on the "modified Intent-to-Treat" population: subjects randomized to receive treatment and treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects Randomized to Receive VOLBELLA® | Subjects Randomized to Receive Restylane-L® | Total
Number analyzed (Participants) | 139 | 141 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (11.94) | 48.3 (12.61) | 47.7 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 139 | 274
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  France | 48 | 49 | 97
  United Kingdom | 91 | 92 | 183

OUTCOME MEASURES:

1. Primary Outcome: Month 3 Overall Lip Fullness Scale Responder Rate Based on Independent Central Reviewer's Assessment
Description: The primary effectiveness variable is the responder rate (percentage of subjects who show ≥ 1-point improvement on the 5-point Lip Fullness Scale (Minimal, Mild, Moderate, Marked, Very Marked) compared to baseline assessment, as determined by Independent Central Reviewer evaluation of 3D photographic images).
Time Frame: 3 months
Population: Per-protocol population (all subjects who are randomized, received at least 1 study treatment, and have no protocol deviations that affect the primary effectiveness endpoint)
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Subjects Randomized to Receive VOLBELLA® and Treated | Subjects Randomized to Receive Restylane-L® and Treated
Number analyzed (Participants) | 123 | 123
Percentage of subjects | 34.1 [25.77 to 42.53] | 29.3 [21.23 to 37.31]
Statistical Analysis 1: Comparison: Subjects Randomized to Receive VOLBELLA® and Treated vs Subjects Randomized to Receive Restylane-L® and Treated; The null hypothesis is that VOLBELLA® is inferior to Restylane-L® in terms of responder rate at Month 3, and the alternative hypothesis is that VOLBELLA® is inferior to Restylane-L® in terms of responder rate at Month 3 with 15% pre-defined non-inferiority margin. To test the null hypothesis, a difference in responder rates of these products (VOLBELLA® - Restylane-L®) at Month 3 and a 1-sided 97.5% Wald confidence interval for the difference is calculated; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is pre-defined as 15% i.e., if the difference in responder rates is significantly greater than -15% (i.e., the lower confidence limit is greater than -15%), statistical non-inferiority of VOLBELLA® to Restylane-L® is established; Difference in responder rates = 4.9, 97.5% CI 1-sided [lower limit -6.7] — Difference in responder rates is calculated as the responder rate at Month 3 for VOLBELLA® minus the responder rate at Month 3 for Restylane-L®

ADVERSE EVENTS:
Arm/Group | Subjects Treated With VOLBELLA® | Subjects Treated With Restylane-L®
Serious Adverse Events (participants affected / at risk) | 1/139 | 1/141
Other Adverse Events (participants affected / at risk) | 27/139 | 26/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Treated With VOLBELLA® (N=139) | Subjects Treated With Restylane-L® (N=141)
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 — This event was classified as not related to the anesthesia, study device, or procedure, and resolved without sequelae after treatment with medication and a procedure.
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — This event was classified as not related to the anesthesia, study device, or procedure, and resolved with sequelae after treatment with a procedure.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Treated With VOLBELLA® (N=139) | Subjects Treated With Restylane-L® (N=141)
Injection site mass (General disorders) | 14 | 12 — lumps/bumps
Injection site pain (General disorders) | 5 | 9
Oral herpes (Infections and infestations) | 11 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Allergan, as the Sponsor, has proprietary interest in this study. Authorship and manuscript composition will reflect joint cooperation between multiple Investigators and sites and Allergan personnel. Authorship will be established prior to the writing of the manuscript. As this study involves multiple centers, no individual publications will be allowed prior to completion of the final report of the multicenter study except as agreed with Allergan.